CLINICAL TRIAL: NCT00275054
Title: Randomized Phase III Trial Comparing Early Treatment With Fludarabine/Cyclophosphamide + Rituximab Versus Deferred Treatment in Untreated Binet Stage A Patients With CLL and High Risk of Progression
Brief Title: Rituximab, Fludarabine, and Cyclophosphamide or Observation Alone in Treating Patients With Stage 0, Stage I, or Stage II Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLL7; EU-20559; ROCHE-GCLLSG-CLL7; 2005-003018-14 (EudraCT Number)
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: stage 0 chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; Cyclophosphamide; Rituximab

ARMS (3):
- Cohort I (FCR) (Experimental): Patients with 2 or more risk factors out of 4 (1. unfavorable molecular cytogenetics, 2. high serum thymidine kinase levels, 3. lymphocyte doubling time shorter than 12 months, 4. unmutated IgVH gene) who are randomized into cohort I receive Fludarabine, Cyclophosphamide and Rituximab (FCR) chemoimmunotherapy.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Rituximab
- Cohort II (W&W) (No Intervention): Patients with 2 or more risk factors out of 4 (1. unfavorable molecular cytogenetics, 2. high serum thymidine kinase levels, 3. lymphocyte doubling time shorter than 12 months, 4. unmutated IgVH gene) who are randomized into cohort II receive no treatment at all (watch & wait).
- Cohort III (W&W) (No Intervention): Patients with less than 2 risk factors out of 4 (1. unfavorable molecular cytogenetics, 2. high serum thymidine kinase levels, 3. lymphocyte doubling time shorter than 12 months, 4. unmutated IgVH gene) are assigned directly to cohort III and receive no treatment at all (watch & wait).

INTERVENTIONS:
Drug: Fludarabine — cycles 1-6: 25 mg/m² i.v., d2-4, q28d
  Other Names: Fludura
  Arms: Cohort I (FCR)
Drug: Cyclophosphamide — cycles 1-6: 250 mg/m² i.v., d2-4, q28d
  Other Names: Endoxan
  Arms: Cohort I (FCR)
Biological: Rituximab — cycle1: 375 mg/m² i.v., d1, q28d
  cycles 2-6: 500 mg/m² i.v., d1, q28d
  Other Names: Mabthera; Rituxan
  Arms: Cohort I (FCR)

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as fludarabine and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Sometimes the cancer may not need treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether giving rituximab together with fludarabine and cyclophosphamide is more effective than observation alone in treating chronic lymphocytic leukemia.

PURPOSE: This randomized phase III trial is studying rituximab, fludarabine, and cyclophosphamide to see how well they work compared to observation alone in treating patients with stage 0, stage I, or stage II B-cell chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effect, in terms of event-free survival, of deferred versus immediate treatment with rituximab, fludarabine, and cyclophosphamide in patients with previously untreated Binet stage A chronic lymphocytic leukemia at high risk for disease progression.
* Investigate and define a new prognostic staging system for patients with Binet stage A chronic lymphocytic leukemia.

Secondary

* Compare the time to progression to Binet stages B and C in patients treated with these regimens.
* Compare the overall and progression-free survival of patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.
* Compare the time to treatment in patients treated with these regimens.
* Analyze the pharmacoeconomics of these regimens in these patients.
* Determine the overall response rate (partial and complete) in patients included in the early treatment arm.
* For patients included in the early treatment arm in complete remission, determine the percentage achieving complete molecular remission using the clone-specific CDR-III region as follow-up parameter.
* Determine the duration of response in patients included in the early treatment arm.
* Determine any adverse events related to treatment/safety of treatment.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to risk factor profile (< 2 risk factors [low risk] vs ≥ 2 risk factors [high risk]). Low-risk patients are assigned to arm II. High-risk patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive rituximab IV on day 1, fludarabine IV on days 1-3, and cyclophosphamide IV on days 1-3. Treatment repeats every 28 days for up to 6 courses.
* Arm II: Patients undergo observation only until disease progression.

PROJECTED ACCRUAL: A total of 600 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Established diagnosis of B-cell chronic lymphocytic leukemia

  * First diagnosis within 12 months before inclusion in study
  * Previously untreated disease
* Binet stage A disease (Rai stage 0, I, or II)

PATIENT CHARACTERISTICS:

* Life expectancy > 6 months
* ECOG performance status 0-2
* Willingness to accept contraception (if randomized to arm I) for the duration of therapy and 12 months thereafter
* Negative serum pregnancy test
* All parameters for risk stratification (lymphocyte doubling time, cytogenetics, unmutated IgVH, and serum thymidine kinase level > 10) present

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiotherapy, or antibody treatment
* No other concurrent chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825 (Actual)
Dates: Start 2005-10; Primary Completion 2007-07 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Event-free survival
Development of a new prognostic staging system

SECONDARY OUTCOMES:
Progression free survival
Overall survival
Time to progression to Binet stages B and C
Time to treatment
Quality of life
Pharmacoeconomic analysis
Overall response (complete and partial) rate in patients in the early treatment arm
Percentage of patients achieving complete molecular remission in the early treatment arm
Duration of response in patients in the early treatment arm
Adverse events in patients in the early treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hallek, MD, Principal Investigator — Medizinische Universitaetsklinik I at the University of Cologne
Locations (91):
- Universitaetsklinik fuer Innere Medizin I, Vienna, Austria
- France (25):
  - Centre Hospitalier Universitaire d'Amiens, Amiens
  - Centre Hospitalier Regional et Universitaire d'Angers, Angers
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Hopital Avicenne, Bobigny
  - CHU de Caen, Caen
  - CHR Clermont Ferrand, Hotel Dieu, Clermont-Ferrand
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Centre Jean Bernard, Le Mans
  - Centre Hospital Universitaire Hop Huriez, Lille
  - Hopital Edouard Herriot - Lyon, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - CHR Hotel Dieu, Nantes
  - Hopital Saint-Louis, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Necker, Paris
  - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - CHU - Robert Debre, Reims
  - Centre Henri Becquerel, Rouen
  - Hopital Universitaire Hautepierre, Strasbourg
  - CHU de Toulouse, Hotel Dieu, Toulouse
  - CHU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (65):
  - Praxis fuer Innere Medizin Haematologie und Internistische Onkologie, Alsfeld
  - Hamatologische/Onkologische Gemeinschaftspraxis - Augsburg, Augsburg
  - Kreiskrankenhaus Aurich, Aurich
  - Klinikum am Bamberg, Bamberg
  - Internistische Gemeinschaftspraxis - Berlin, Berlin
  - St. Hedwig Krankenhaus, Berlin
  - Internistische Gemeinschaftspraxis Betzdorf, Betzdorf
  - DIAKO Ev. Diakonie Krankenhaus gGmbH, Bremen
  - Onkologische Schwerpunktpraxis at Facharzt fuer Innere Medizin, Coesfeld
  - Praxis Fuer Haematologie Internistische Onkologie, Cologne
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Helios Klinikum Erfurt, Erfurt
  - Onkologische Schwerpunkt Praxis, Erlangen
  - St. Antonius Hospital, Eschweiler
  - Universitaetsklinikum Essen, Essen
  - Internistische Gemeinschaftspraxis - Forchheim, Forchheim
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Internistische Gemeinschaftspraxis - Friedberg, Friedberg
  - Fürstenzell
  - Klinikum Garmisch - Partenkirchen GmbH, Garmisch-Partenkirchen
  - Internistische Praxisgemeinschaft, Germering
  - Gemeinschaftspraxis Fuer Innere Medizin, Hematologie Und Onkologie, Giessen
  - Universitaetsklinikum Goettingen, Göttingen
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Maria-Josef-Hospital Greven GmbH, Greven
  - St. Marien Hospital - Katholisches Krankenhaus Hagen gGmbH, Hagen
  - Internistische Gemeinschaftspraxis - Halle, Halle
  - Universitaetsklinikum Halle, Halle
  - Krankenhaus Siloah - Medizinische Klinik II, Hanover
  - Praxis Dr. med Freddy Henne, Hechingen
  - Universitatsklinikum Heidelberg, Heidelberg
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Internistische Gemeinschaftspraxis - Kassel, Kassel
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Internistische Onkologische Praxis - Kronach, Kronach
  - Internistische Praxis - Landshut, Landshut
  - Caritas - Krakenhaus Lebach, Lebach
  - Onkologische Schwerpunktpraxis - Leer, Leer
  - Staedtisches Klinikum Magdeburg - Altstadt, Magdeburg
  - Gemeinschaftspraxis, Mannheim
  - Klinikum Minden, Minden
  - Monchenglasbach/Rheydt
  - Haematologische Praxis - Moenchengladbach, Mönchengladbach
  - Munich Oncologic Practice at Elisenhof, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Hamatologie/Onkologie Praxisgemeinschaft - Muenchen, Munich
  - Haematologische Schwerpunktpraxis, Munich
  - Klinikum Schwaebisch Gmuend Stauferklinik, Mutlangen
  - Internistische Gemeinschaftspraxis - Offenbach, Offenbach
  - Internistische Gemeinschaftspraxis - Oldenburg, Oldenburg
  - Pforzheim
  - Internistische Schwerpunktpraxis, Rüsselsheim am Main
  - Schwerpunktpraxis fuer Haematologie und Onkologie, Saarbrücken
  - Diakonie - Krankenhaus, Schwäbisch Hall
  - St. Marien - Krankenhaus Siegen GMBH, Siegen
  - Singen
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Diakonie Klinikum Stuttgart, Stuttgart
  - Onkologische Gemeinschaftspraxis - Trier, Trier
  - Universitaetsklinikum Tuebingen, Tübingen
  - Praxis fuer Haematologie und Onkologie, Twistringen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - St. Marienhospital - Vechta, Vechta
  - Burkhard and Reimann Gemeinschaftspraxis, Worms

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sachanas S, Pangalis GA, Fink AM, Bahlo J, Fischer K, Levidou G, Kyrtsonis MC, Bartzi V, Vassilakopoulos TP, Kalpadakis C, Koulieris E, Moschogiannis M, Yiakoumis X, Tsirkinidis P, Angelopoulou MK, Eichhorst B, Hallek M. Small Lymphocytic Lymphoma: Analysis of Two Cohorts Including Patients in Clinical Trials of the German Chronic Lymphocytic Leukemia Study Group (GCLLSG) or in "Real-Life" Outside of Clinical Trials. Anticancer Res. 2019 May;39(5):2591-2598. doi: 10.21873/anticanres.13382. PMID 31092457
- [Derived] Herling CD, Cymbalista F, Gross-Ophoff-Muller C, Bahlo J, Robrecht S, Langerbeins P, Fink AM, Al-Sawaf O, Busch R, Porcher R, Cazin B, Dreyfus B, Ibach S, Lepretre S, Fischer K, Kaiser F, Eichhorst B, Wentner CM, Hoechstetter MA, Dohner H, Leblond V, Kneba M, Letestu R, Bottcher S, Stilgenbauer S, Hallek M, Levy V. Early treatment with FCR versus watch and wait in patients with stage Binet A high-risk chronic lymphocytic leukemia (CLL): a randomized phase 3 trial. Leukemia. 2020 Aug;34(8):2038-2050. doi: 10.1038/s41375-020-0747-7. Epub 2020 Feb 18. PMID 32071431